CLINICAL TRIAL: NCT02283671
Title: Treatment of Multiple Sclerosis and Neuromyelitis Optica With Regulatory Dendritic Cell: Clinical Trial Phase 1 B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sara Varea (Other)
Responsible Party: Sponsor-Investigator, Sara Varea, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TolDec-EM-NMO
Record Dates: First submitted 2014-10-29; First posted 2014-11-05 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis; Neuromyelitis Optica
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tolerogenic dendritic cells (Experimental): Somatic-cell therapy medicines: tolerogenic dendritic cells loaded with myelin peptides.
  Patients will receive intravenous administration every two weeks (week 0 , 2 and 4 ) representing a total of three administrations per patient.
  The dose escalation will occur as expected in the absence of limiting toxicity in the previous dosage level.
  Interventions: Biological: Tolerogenic Dendritic cells loaded with myelin peptides

INTERVENTIONS:
Biological: Tolerogenic Dendritic cells loaded with myelin peptides — Somatic-cell therapy medicines application

SUMMARY:
First in human study to assess the tolerability and safety profile of treatment with dendritic cell in patients with multiple sclerosis or neuromyelitis optica.

ELIGIBILITY:
Inclusion Criteria:

* patients with Multiple sclerosis or neuromyelitis optica
* diagnosed more than a year before inclusion
* Expanded Disability Status Scale between 3.0 and 8.5
* all subtypes of multiple sclerosis or Neuromyelitis optica
* Multiple Sclerosis patients who have previously been offered therapeutic alternatives available in indications and either decline or that after receiving treatment for at least 6 months have had an outbreak or an increase of at least 1 point on the Expanded Disability Status Scale (EDSS) (non-responders) or who have not tolerated treatment
* Patients with Neuromyelitis optica (NMO) in stable immunomodulatory treatment in the past 6 months or without treatment because they are not candidates to receive it

Exclusion Criteria:

* Corticosteroid treatment in the last 30 days
* Presence of an outbreak in the last month
* Inability to perform brain Magnetic resonance imaging (with paramagnetic contrast)
* Serious systemic diseases, including Hepatitis B virus, Hepatitis C Virus, and Human Immunodeficiency Virus. Uncontrolled hypertension, insulin-dependent diabetes mellitus, heart disease or kidney failure or severe respiratory
* Personal history of cancer or family history of known hereditary cancer
* patient participating in other experimental study in the last 3 months
* women childbearing-aged that do not use effective contraceptive methods
* pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
number of patients with adverse events | after 12 weeks of follow up

SECONDARY OUTCOMES:
Multiple Sclerosis Functional Composite scale | after 12 weeks of follow up
Multiple Sclerosis Spasticity Scale | after 12 weeks of follow up
Expanded Disability Status Scale | after 12 weeks of follow up
SF36 Health Status questionnaire | after 12 weeks of follow up
EuroQol5D | after 12 weeks of follow up
Changes in immunological profile | after 12 weeks of follow up
number of disease outbreaks | after 12 weeks of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Villoslada, MD PhD, Study Chair — Institut d'Investigacions Biomèdiques August Pi i Sunyer
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain